CLINICAL TRIAL: NCT05693831
Title: myCare-102: A Survey of Physician and Molecular Tumor Board Perspectives on the Clinical Utility and Usability of Cellworks Singula™ and Cellworks Ventura™ Reports in Facilitating Patient Treatment Decisions for Pan-Cancer Patients
Brief Title: myCare-102: Clinical Utility and Usability of Cellworks Singula™ and Cellworks Ventura™ Reports
Acronym: myCare-102
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cellworks Group Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: myCare-102
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Cancer; Relapsed Cancer; Refractory Cancer
Keywords: cancer; relapsed/refractory; second-line therapy; third-line therapy; received first-line therapy
MeSH Terms: conditions — Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Singula: Patients with a diagnosis of cancer who have already received first line therapy
  Interventions: Other: Cellworks Report
- Ventura: Patients with a diagnosis of relapsed or refractory cancer
  Interventions: Other: Cellworks Report

INTERVENTIONS:
Other: Cellworks Report — Survey physicians and molecular tumor board perspectives of the benefit of Cellworks Singula™ and Ventura™ reports in facilitating treatment decisions in pan-cancer patients.
  Other Names: Cellworks Singula Report; Cellworks Ventura Report

SUMMARY:
The purpose of this study is to determine the benefit of Cellworks Singula™ reports on physician and molecular tumor board treatment recommendations across a large set of pan-cancer indications who have already received first-line therapy. The study is also to determine the benefit of Cellworks Ventura™ reports on physician and molecular tumor board treatment recommendations across a large set of relapsed or refractory pan-cancer indications.

The primary objective of this study is to survey physicians and molecular tumor board perspectives of the benefit of Cellworks Singula™and Cellworks Ventura™ reports in facilitating treatment decisions in pan-cancer patients.

Cellworks reports aim to provide NGS-based therapy recommendations to aid the decision-making of patients, physicians, and molecular tumor boards. Cellworks reports aim to provide NGS-based therapy recommendations to aid the decision-making of patients, physicians, and molecular tumor boards.

ELIGIBILITY:
Inclusion Criteria:

* Have cancer for the indications listed at: https://cellworks.life/mycare102. Patients are eligible at any stage of the disease.
* Have already received first-line therapy
* For Cellworks Singula™ report, patients must be Relapsed or refractory after first-line treatment.
* For Cellworks Ventura™ report, patients must have relapsed or refractory cancer and have exhausted standard of care therapy options
* Expected to be alive 6 months or more
* Requirements for NGS testing (e.g., panel or whole-exome sequencing)
* NGS testing has been ordered from or performed by one or more vendors specified at: https://cellworks.life/mycare102
* NGS reports must be ordered or performed within the last 90 days
* Cellworks will accept all NGS input formats available, including PDF, VCF, BAM, and FastQ.
* Requirements for additional laboratory testing: If Hematological Indication then Cytogenetics in the form of FISH, Karyotyping, IHC, and/or aCGH has been ordered. If Acute Myeloid Leukemia (AML) then FLT3-itd testing has been ordered. If the Indication is a form of Brain Cancer (e.g., glioblastoma) then Cytogenetics in the form of FISH, Karyotyping, IHC, and/or aCGH has been ordered and MGMT Methylation test has been ordered.

Exclusion Criteria:

* Patients not previously diagnosed with cancer of any of the indications listed at: https://cellworks.life/mycare102
* Patients without an NGS report ordered/performed within the past 90 days
* Patients who are expected to be alive less than 6 months
* Pregnant women
* Patients who have not exhausted standard-of-care treatment options or who have known effective therapy
* Patients that fall into the following categories based on survey response will considered excluded from eligibility: If recommendations were made before receiving the Cellworks report, patients will not be included in the primary analysis but will be included in the ITT analysis. If recommended an FDA approved therapy that was not included on the Cellworks report. If recommended a clinical trial for a therapy that was not included in the Cellworks report. If the therapy/therapies on the Cellworks report was/were not covered by the patient's insurance. If the therapy/therapies on the Cellworks report was/were too expensive.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients with a diagnosis of cancer who have already received first line therapy, for Cellworks Singula™ report.
  * Patients with a diagnosis of relapsed or refractory cancer, for Cellworks Ventura™ report.
Sampling Method: Non-Probability Sample
Enrollment: 730 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Surveyed View of Cellworks Singula and Ventura™ reports | Approximately 24 months
  Majority of physicians and molecular tumor boards (MTB) have a positive view of the Cellworks Singula™ and Cellworks Ventura™ reports

SECONDARY OUTCOMES:
Patient Demographics (Sex) | Approximately 24 months
  Patient Sex
Patient Demographics (Ethnicity) | Approximately 24 months
  Ethnicity
Patient Demographics (Age) | Approximately 24 months
  Age
Institution Demographics (Type) | Approximately 24 months
  Institution Type
Institution Demographics (Orders Placed) | Approximately 24 months
  Number of Orders Placed
Institution Demographics (Placement of Orders) | Approximately 24 months
  Placement Within Orders
Patient Disease Status (Indication) | Approximately 24 months
  Disease Indication
Patient Disease Status (ECOG) | Approximately 24 months
  ECOG Score

CONTACTS AND LOCATIONS:
Overall Officials: Scott Howard, M.D., Principal Investigator — University of TN Health Science Center; Tobias Meissner, Dr. sc. hum., Principal Investigator — Avera Cancer Institute
Locations (1):
- Avera Cancer Institute, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No